CLINICAL TRIAL: NCT03108365
Title: Evaluating the Effectiveness of Axiostat Hemostatic Dressing Material Versus Conventional Method of Hemostasis and Healing of Extraction Wounds in Patients on Oral Anti-Platelet Drugs - A Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Axio Biosolutions Pvt. Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABPL/004
Record Dates: First submitted 2017-03-30; First posted 2017-04-11 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2017-04

CONDITIONS: Tooth Extraction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Axiostat (Experimental): Size: 1 x 1 cm
  Chitosan based haemostatic dressing
  Interventions: Device: Axiostat
- Cotton Gauze (Active Comparator): Size: 1 x 1 cm
  Interventions: Device: Cotton Gauze

INTERVENTIONS:
Device: Axiostat — Axiostat® is a sterile, non-absorbable haemostatic dressing intended to control profuse bleeding within minutes of application by providing an active mechanical barrier to the wound site.
  Axiostat® stops moderate to severe bleeding due to cuts, abrasions, lacerations, venous/arterial punctures and more. Mechanism of action is such that Axiostat® is an extremely positive dressing that becomes very sticky in the presence of negatively charged blood and thus seals the wound area.
  Other Names: Chitosan haemostatic dressing
  Arms: Axiostat
Device: Cotton Gauze — Size: 1 x 1 cm
  Arms: Cotton Gauze

SUMMARY:
The rationale of this study was to evaluate the efficacy of Axiostat hemostatic dental dressing in achieving hemostasis post-extraction and determining its effect on pain and healing of the extraction wound, compared to control, i.e. conventional method of extraction in patients on oral anti-platelet therapy.

ELIGIBILITY:
Inclusion criteria

* Patients undergoing multiple tooth extractions aged b/w 35- 70 years and with INR values ≤ 3.5 (1-3.5)
* If present, sugar level should be under control

Exclusion criteria

* Patients undergoing a single tooth or multiple extractions in same quadrant; and those with an allergy to seafood.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-12-19 (Actual); Primary Completion 2016-03-24 (Actual); Study Completion 2016-03-24 (Actual)

PRIMARY OUTCOMES:
Time to achieve haemostasis | 1 Day
  Time to achieve hemostasis by observing the time at which blood oozing through or from periphery of the dressing stops.

SECONDARY OUTCOMES:
Pain & Healing Scale | Upto 1 Day
  Patients comfort level as assessed by verbal inquiry after completion of procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Tejraj Kale, Principal Investigator — KLE Dental College, Belgaun

REFERENCES:
- See also: Publication in Journal of Contemporary Dental Medicine — https://www.ncbi.nlm.nih.gov/pubmed/?term=Axiostat